CLINICAL TRIAL: NCT01421459
Title: A Prospective, Randomized, Double-Blind Comparison of a Long-Acting Basal Insulin Analog LY2963016 to Lantus in Adult Patients With Type 2 Diabetes Mellitus: The ELEMENT 2 Study
Brief Title: A Study in Adults With Type 2 Diabetes
Acronym: ELEMENT 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13713; I4L-MC-ABEC (Other: Eli Lilly and Company); 2011-000828-15 (EudraCT Number)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2963016 + OAMs (Experimental): LY2963016 titrated based on blood glucose readings, administered subcutaneously, once daily in combination with at least 2 oral antihyperglycemic medications (OAMs) [alpha glucosidase inhibitors (AGI), dipeptidyl peptidases intravenous (DPP-IV), meglitinide (MEG), metformin (MET), sulfonylurea (SU), and thiazolidinedione (TZD)] administered per standard of care for 24 weeks
  Interventions: Drug: LY2963016; Drug: OAMs
- Lantus + OAMs (Active Comparator): Lantus titrated based on blood glucose readings, administered subcutaneously, once daily in combination with at least 2 OAMs (AGI, DPP-IV, MEG, MET, SU, and TZD) administered per standard of care for 24 weeks
  Interventions: Drug: Lantus; Drug: OAMs

INTERVENTIONS:
Drug: LY2963016 — Administered subcutaneously
  Arms: LY2963016 + OAMs
Drug: Lantus — Administered subcutaneously
  Arms: Lantus + OAMs
Drug: OAMs — Administered orally

SUMMARY:
The main purpose of this study is to compare the effectiveness and safety of LY2963016 versus Lantus in controlling blood sugar levels in combination with two or more oral diabetes medications.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes Mellitus based on the disease diagnostic criteria World Health Organization (WHO) classification
* Have been taking at least 2 types of oral diabetes medications for at least 12 weeks prior to entering the study
* Have a Hemoglobin A1c value greater than or equal to 7.0 percent and less than or equal to 11.0 percent if insulin naive If previously on Lantus, then Hemoglobin A1c must be less than or equal to 11.0 percent
* Have a body mass index of less than or equal to 45 kilogram per meter squared (kg/m^2)

Exclusion Criteria:

* Have significant liver, cardiac or gastrointestinal disease
* Have active cancer or have had cancer within the past 5 years (with the exception of basal cell carcinoma or carcinoma in situ)
* Have an excessive resistance to insulin or hypersensitivity to Lantus
* Have had more than one episode of severe low blood sugar (defined as needing someone else to help because you had very low blood sugar) within the 6 months before entering the study
* Have taken any other insulin other than Lantus within the past 30 days
* Taking any other diabetes medicines that are not allowed in the study or not approved to be taken with insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (62):
- United States (28):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montgomery, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooksville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roswell, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Gibson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mineola, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hurst, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longview, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plano, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandýs nad Labem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vieux-Condé
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aschaffenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giengen an der Brenz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lüneburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Ingbert-Oberwürzbach
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki, Greece
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pápa
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara Jalisco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ruda Śląska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yong Kung City

REFERENCES:
- [Derived] Nishiyama H, Shingaki T, Suzuki Y, Ilag LL. Similar Intrapatient Blood Glucose Variability with LY2963016 and Lantus(R) Insulin Glargine in Patients with Type 1 (T1D) or Type 2 Diabetes, Including a Japanese T1D Subpopulation. Diabetes Ther. 2018 Aug;9(4):1469-1476. doi: 10.1007/s13300-018-0450-0. Epub 2018 May 31. PMID 29855972
- [Derived] Pollom RK, Costigan T, Lacaya LB, Ilag LL, Hollander PA. Similar Efficacy and Safety of Basaglar(R) and Lantus(R) in Patients with Type 2 Diabetes in Age Groups (< 65 Years, >/= 65 Years): A Post Hoc Analysis from the ELEMENT-2 Study. Diabetes Ther. 2018 Apr;9(2):827-837. doi: 10.1007/s13300-018-0405-5. Epub 2018 Mar 14. PMID 29542012

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2963016 + OAMs: LY2963016 titrated based on blood glucose (BG) readings, administered subcutaneously, once daily in combination with at least 2 oral antihyperglycemic medications (OAMs) administered per standard of care for 24 weeks
- Lantus + OAMs: Lantus titrated based on BG readings, administered subcutaneously, once daily in combination with at least 2 OAMs administered per standard of care for 24 weeks
Period: Overall Study
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Started | 379 | 380
Received at Least 1 Dose of Study Drug | 376 | 380
Completed | 334 | 328
Not Completed | 45 | 52
Not completed — Adverse Event | 6 | 10
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 8 | 9
Not completed — Physician Decision | 9 | 9
Not completed — Protocol Violation | 8 | 5
Not completed — Withdrawal by Subject | 12 | 16

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2963016 + OAMs | Lantus + OAMs | Total
Number analyzed (Participants) | 376 | 380 | 756
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.98 (10.17) | 58.67 (10.02) | 58.82 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 181 | 378
  Male | 179 | 199 | 378
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 106 | 104 | 210
  Not Hispanic or Latino | 244 | 256 | 500
  Unknown or Not Reported | 26 | 20 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 21 | 38
  Asian | 29 | 35 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 32 | 58
  White | 302 | 291 | 593
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czech Republic | 18 | 18 | 36
  France | 8 | 8 | 16
  Germany | 15 | 13 | 28
  Greece | 10 | 12 | 22
  Hungary | 32 | 30 | 62
  Italy | 6 | 5 | 11
  Korea, Republic of | 17 | 15 | 32
  Mexico | 29 | 29 | 58
  Poland | 12 | 11 | 23
  Puerto Rico | 39 | 31 | 70
  Spain | 10 | 12 | 22
  Taiwan | 9 | 12 | 21
  United States | 171 | 184 | 355
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  percentage of glycosylated hemoglobin | 8.34 (1.09) | 8.31 (1.06) | 8.33 (1.08)
Sulfonylurea Use [Number; unit: participants] — Number of participants who used or did not use sulfonylurea.
  participants
    Yes, did use sulfonylurea | 315 | 315 | 630
    No, did not use sulfonylurea | 61 | 65 | 126
Time of Basal Insulin Injection [Number; unit: participants] — Number of participants who administered a basal insulin injection during the Daytime and Evening/Bedtime.
  participants
    Daytime | 187 | 188 | 375
    Evening/Bedtime | 189 | 192 | 381
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 90.35 (20.02) | 89.83 (19.25) | 90.09 (19.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline up to 24 Weeks in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection and treatment.
Time Frame: Baseline, Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug and with a Baseline and at least 1 post-Baseline HbA1c measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 369 | 375
percentage of glycosylated hemoglobin | -1.286 (0.06) | -1.338 (0.06)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Non-Inferiority or Equivalence — The primary treatment comparison was to compare LY2963016 versus Lantus at the non-inferiority margin of +0.4%. If the upper limit of the 95% confidence interval on the change from baseline to 24-week endpoint HbA1c for LY2963016 versus Lantus was below +0.4%, then LY2963016 would be declared non-inferior to Lantus; p = 0.403, ANCOVA; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.070 to 0.175]

2. Secondary Outcome: Change From Baseline in Insulin Antibody Levels
Description: Blood samples are collected from participants and percentage of insulin antibody binding measured. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline of response and treatment.
Time Frame: Baseline and 4 weeks and 12 weeks and Endpoint (24 weeks and up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug and with a Baseline and at least 1 post-Baseline insulin antibody measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of insulin antibody binding
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 14 | 6
percentage of insulin antibody binding
  Change at 4 weeks (n=10, 3) | -1.07 (1.47) | -3.25 (2.79)
  Change at 12 weeks (n=9, 5) | -1.57 (1.14) | -4.39 (1.54)
  Change at 24 weeks (n=10, 2) | -2.61 (0.60) | -3.21 (1.35)
  Change at Endpoint, up to 24 weeks (n=14, 6) | -2.49 (0.39) | -3.11 (0.06)

3. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection and treatment.
Time Frame: Baseline and 4 weeks and 8 weeks and 12 weeks and 16 weeks and 20 weeks and 24 weeks
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline HbA1c measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 369 | 375
percentage of HbA1c
  Change at 4 weeks (n=368, 371) | -0.452 (0.03) | -0.481 (0.03)
  Change at 8 weeks (n=359, 358) | -0.871 (0.05) | -0.866 (0.05)
  Change at 12 weeks (n=349, 351) | -1.134 (0.06) | -1.143 (0.06)
  Change at 16 weeks (n=345, 345) | -1.265 (0.06) | -1.321 (0.06)
  Change at 20 weeks (n=338, 334) | -1.294 (0.06) | -1.379 (0.06)
  Change at 24 weeks (n=331, 329) | -1.336 (0.06) | -1.438 (0.06)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.382, ANCOVA — P-value is for 4 weeks
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.910, ANCOVA — P-value is for 8 weeks
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.869, ANCOVA — P-value is for 12 weeks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.345, ANCOVA — P-value is for 16 weeks
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.161, ANCOVA — P-value is for 20 weeks
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.097, ANCOVA — P-value is for 24 weeks

4. Secondary Outcome: 7-Point Self-Monitored Blood Glucose (SMBG) Profiles
Description: Seven-point SMBG are completed at the following timepoints: Morning (AM) Pre-Meal, Morning (AM) Post-Prandial (PP), Midday (MD) Pre-Meal, Midday PP, Evening (EV) Pre-Meal, Bed Time and 0300 hours. PP glucose is measured 2 hours (hrs) after the start of the meal. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection, and treatment.
Time Frame: Baseline and Endpoint [up to 24 weeks (wk)]
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline SMBG measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 357 | 359
millimoles per liter (mmol/L)
  Baseline- AM Pre-Meal (n=353, 359) | 8.82 (0.13) | 8.86 (0.13)
  Baseline- AM 2 hrs PP (n=356, 356) | 11.68 (0.16) | 11.80 (0.16)
  Baseline- MD Pre-Meal (n=357, 357) | 9.09 (0.15) | 9.44 (0.15)
  Baseline- MD 2 hrs PP (n=357, 353) | 10.65 (0.15) | 10.89 (0.15)
  Baseline- EV Pre-Meal (n=356, 354) | 9.29 (0.15) | 9.59 (0.15)
  Baseline- Bed Time (n=355, 354) | 11.25 (0.16) | 11.17 (0.16)
  Baseline- 0300 hrs (n=342, 341) | 8.83 (0.15) | 8.96 (0.15)
  Endpoint, up to 24 wk- AM Pre-Meal (n=353, 359) | 5.94 (0.11) | 6.06 (0.11)
  Endpoint, up to 24 wk- AM 2 hrs PP (n=356, 356) | 8.07 (0.17) | 8.40 (0.17)
  Endpoint, up to 24 wk- MD Pre-Meal (n=357, 357) | 6.81 (0.15) | 7.12 (0.15)
  Endpoint, up to 24 wk- MD 2 hrs PP (n=357, 353) | 8.53 (0.17) | 8.69 (0.18)
  Endpoint, up to 24 wk- EV Pre-Meal (n=356, 354) | 7.29 (0.16) | 7.40 (0.16)
  Endpoint, up to 24 wk- Bed Time (n=355, 354) | 8.56 (0.18) | 8.67 (0.18)
  Endpoint, up to 24 wk- 0300 hrs (n=342, 341) | 6.72 (0.15) | 6.70 (0.15)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.837, ANCOVA — P-value is at Morning Pre-Meal at Baseline
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.620, ANCOVA — P-value is for Morning 2 hrs PP Meal at Baseline
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.107, ANCOVA — P-value is for Midday Pre-Meal at Baseline
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.258, ANCOVA — P-value is for Midday 2 hrs PP Meal at Baseline
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.161, ANCOVA — P-value is for Evening Pre-Meal at Baseline
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.725, ANCOVA — P-value is for Bed Time at Baseline
Statistical Analysis 7: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.543, ANCOVA — P-value is for 0300 hrs at Baseline
Statistical Analysis 8: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.265, ANCOVA — P-value is for Morning Pre-Meal at Endpoint, up to 24 wk
Statistical Analysis 9: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.050, ANCOVA — P-value is for Morning 2 hrs PP Meal at Endpoint, up to 24 weeks
Statistical Analysis 10: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.040, ANCOVA — P-value is for Midday Pre-Meal at Endpoint, up to 24 weeks
Statistical Analysis 11: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.366, ANCOVA — P-value is for Midday 2 hrs PP Meal at Endpoint, up to 24 weeks
Statistical Analysis 12: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.485, ANCOVA — P-value is for Evening Pre-Meal at Endpoint, up to 24 weeks
Statistical Analysis 13: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.537, ANCOVA — P-value is for Bed Time at Endpoint, up to 24 weeks
Statistical Analysis 14: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.878, ANCOVA — P-value is for 0300 hrs at Endpoint, up to 24 weeks

5. Secondary Outcome: Glycemic Variability of Fasting Blood Glucose
Description: Glycemic variability is measured by the intra-participant standard deviation (SD) value of fasting blood glucose as measured by the actual morning pre-meal blood glucose value from the 7-point self-monitoring blood glucose [SMBG] profiles. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for baseline HbA1c, country, sulfonylurea use, time of basal insulin injection, and treatment.
Time Frame: Baseline and Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline fasting blood glucose measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 342 | 345
millimoles per liter (mmol/L)
  Baseline | 1.18 (0.05) | 1.20 (0.05)
  Endpoint, up to 24 weeks | 0.81 (0.06) | 0.79 (0.06)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.779, ANCOVA — P-value is for Baseline
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.788, ANCOVA — P-value is for Endpoint, up to 24 weeks

6. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection, and treatment.
Time Frame: Baseline and 4 weeks (wk) and 8 wk and 12 wk and 16 wk and 20 wk and 24 wk and Endpoint (up to 24 wk)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline body weight measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 370 | 374
kilogram (kg)
  Change at 4 wk (n=361, 364) | 0.292 (0.11) | 0.526 (0.11)
  Change at 8 wk (n=358, 357) | 0.999 (0.16) | 1.152 (0.16)
  Change at 12 wk (n=350, 352) | 1.271 (0.19) | 1.440 (0.19)
  Change at 16 wk (n=342, 344) | 1.550 (0.22) | 1.918 (0.22)
  Change at 20 wk (n=340, 333) | 1.734 (0.25) | 2.234 (0.25)
  Change at 24 wk (n=335, 329) | 1.914 (0.27) | 2.175 (0.27)
  Change at Endpoint, up to 24 wk (n=370, 374) | 1.776 (0.25) | 2.020 (0.25)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.687, ANCOVA — P-value is for Baseline
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.036, ANCOVA — P-value is for change at 4 wks
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.323, ANCOVA — P-value is for change at 8 wks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.368, ANCOVA — P-value is for change at 12 wks
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.089, ANCOVA — P-value is for change at 16 wks
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.041, ANCOVA — P-value is for change at 20 wks
Statistical Analysis 7: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.330, ANCOVA — P-value is for change at 24 wks
Statistical Analysis 8: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.334, ANCOVA — P-value is for change at Endpoint, up to 24 wks

7. Secondary Outcome: Adult Low Blood Sugar Survey (ALBSS)
Description: ALBSS contains 33 items, with each item scored on a 5-point response scale: 0 (never) to 4 (almost always). Items are categorized in 2 domains: Behavior (or avoidance) Items 1 to 15 and Worry (or affect) Items 16 to 33. Behavior Total Score range is 0 to 60 and Worry Total Score range is 0 to 72. Higher scores on "Behavior" items (related to avoidance of hypoglycemia) reflect greater awareness and/or effort of the participant to prevent low blood sugar. Higher scores on "Worry" items (related to worries about low blood sugar and its consequences) reflect greater participant concern about having low blood sugar. The ALBSS Total Scores (Worry and Behavior item scores combined) range is 0 to 132. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection, and treatment.
Time Frame: 4 weeks (wk) and 12 wk and Endpoint (up to 24 wk)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline ALBSS measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 368 | 371
units on a scale
  Behavior Score- 4 wk (n=351, 354) | 8.41 (0.63) | 8.64 (0.64)
  Behavior Score- 12 wk (n=350, 349) | 8.95 (0.62) | 9.36 (0.62)
  Behavior Score- Endpoint up to 24 wk (n=368, 371) | 7.90 (0.60) | 8.36 (0.60)
  Worry Score- 4 wk (n=352, 354) | 7.74 (0.91) | 8.82 (0.92)
  Worry Score- 12 wk (n=349, 348) | 8.35 (0.91) | 8.51 (0.91)
  Worry Score- Endpoint up to 24 wk (n=368, 371) | 8.61 (0.89) | 8.57 (0.90)
  ALBSS Total Score- 4 wk (n=352, 354) | 16.15 (1.29) | 17.45 (1.29)
  ALBSS Total Score- 12 wk (n=349, 348) | 17.32 (1.32) | 17.85 (1.32)
  ALBSS Total Score-Endpoint up to 24 wk (n=368,371) | 16.53 (1.32) | 16.92 (1.33)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.726, ANCOVA — P-value is for Behavior domain at 4 weeks
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.502, ANCOVA — P-value is for Behavior domain at 12 weeks
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.437, ANCOVA — P-value is for Behavior domain at Endpoint, up to 24 weeks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.237, ANCOVA — P-value is for Worry domain at 4 weeks
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.860, ANCOVA — P-value is for Worry domain at 12 weeks
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.966, ANCOVA — P-value is for Worry domain at Endpoint, up to 24 weeks
Statistical Analysis 7: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.313, ANCOVA — P-value is for ALBSS Total Score at 4 weeks
Statistical Analysis 8: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.683, ANCOVA — P-value is for ALBSS Total Score at 12 weeks
Statistical Analysis 9: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.765, ANCOVA — P-value is for ALBSS Total Score at Endpoint, up to 24 weeks

8. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ)
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. Items divided into 5 domains of satisfaction: Inconvenience of Regimen [(IR) 5 items: domain scores range (DSR) 5-35], Lifestyle Flexibility [(LF) 3 items: DSR 3-21], Glycemic Control [(GC) 3 items: DSR 3-21], Hypoglycemic Control [(HC) 5 items: DSR 5-35], Insulin Delivery Device [(IDD) 6 items: DSR 6-42]. All items measured on a 7-point scale: 1 (no bother at all) to 7 (a tremendous bother), with lower scores reflecting better outcomes. ITSQ Total Overall Raw Scores range from 22-154. Both raw domain and overall scores are transformed on a scale of 0-100, where transformed score=100*[(7-mean raw score)/6]. Higher scores indicate better treatment satisfaction. Least Squares (LS) mean are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection, and treatment.
Time Frame: 4 weeks (wk) and 12 wk and Endpoint (EP) (up to 24 wk)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline ITSQ measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 368 | 372
units on a scale
  IR- 4 wk (n=352, 354) | 86.10 (1.24) | 86.12 (1.25)
  IR- 12 wk (n=350, 348) | 83.44 (1.25) | 84.54 (1.25)
  IR- EP, up to 24 wk (n=368, 371) | 85.62 (1.31) | 85.21 (1.32)
  LF- 4 wk (n=352, 354) | 79.65 (1.55) | 79.87 (1.55)
  LF-12 wk (n=350, 350) | 76.69 (1.52) | 78.16 (1.52)
  LF- EP, up to 24 wk (n=368, 372) | 78.00 (1.51) | 78.32 (1.52)
  HC- 4 wk (n=352, 354) | 79.36 (1.46) | 80.33 (1.46)
  HC- 12 wk (n=350, 348) | 77.15 (1.49) | 77.73 (1.49)
  HC- EP, up to 24 wk (n=368, 372) | 77.51 (1.54) | 79.08 (1.55)
  GC- 4 wk (n=352, 354) | 75.67 (1.62) | 75.47 (1.63)
  GC- 12 wk (n=350, 347) | 78.95 (1.53) | 81.38 (1.53)
  GC- EP, up to 24 wk (n=368, 372) | 80.74 (1.53) | 80.26 (1.54)
  IDD- 4 wk (n=352, 353) | 70.56 (1.56) | 73.22 (1.56)
  IDD- 12 wk (n=348, 349) | 70.97 (1.70) | 72.21 (1.69)
  IDD- EP, up to 24 wk (n=368, 372) | 72.85 (1.63) | 73.87 (1.64)
  ITSQ Overall Total- 4 wk (n=352, 354) | 78.02 (1.12) | 78.98 (1.12)
  ITSQ Overall Total- 12 wk (n=349, 348) | 77.06 (1.21) | 78.30 (1.20)
  ITSQ Overall Total- EP, up to 24 wk (n=368, 372) | 78.54 (1.21) | 79.06 (1.22)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.983, ANCOVA — P-value is for Inconvenience of Regimen at 4 weeks
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.371, ANCOVA — P-value is for Inconvenience of Regimen at 12 weeks
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.757, ANCOVA — P-value is for Inconvenience of Regimen at Endpoint, up to 24 weeks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.890, ANCOVA — P-value is for Lifestyle Flexibility at 4 weeks
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.326, ANCOVA — P-value is for Lifestyle Flexibility at 12 weeks
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.831, ANCOVA — P-value is for Lifestyle Flexibility at Endpoint, up to 24 weeks
Statistical Analysis 7: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.507, ANCOVA — P-value is for Hypoglycemic Control at 4 weeks
Statistical Analysis 8: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.690, ANCOVA — P-value is for Hypoglycemic Control at 12 weeks
Statistical Analysis 9: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.307, ANCOVA — P-value is for Hypoglycemic Control at Endpoint, up to 24 weeks
Statistical Analysis 10: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.902, ANCOVA — P-value is for Glycemic Control at 4 weeks
Statistical Analysis 11: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.109, ANCOVA — P-value is for Glycemic Control at 12 weeks
Statistical Analysis 12: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.754, ANCOVA — P-value is for Glycemic Control at Endpoint, up to 24 weeks
Statistical Analysis 13: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.088, ANCOVA — P-value is for Insulin Deliver Device at 4 weeks
Statistical Analysis 14: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.456, ANCOVA — P-value is for Insulin Delivery Device at 12 weeks
Statistical Analysis 15: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.531, ANCOVA — P-value is for Insulin Delivery Device at Endpoint, up to 24 weeks
Statistical Analysis 16: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.393, ANCOVA — P-value is for ITSQ Total Score at 4 weeks
Statistical Analysis 17: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.296, ANCOVA — P-value is for ITSQ Total Score at 12 weeks
Statistical Analysis 18: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.662, ANCOVA — P-value is for ITSQ Total Score at Endpoint, up to 24 weeks

9. Secondary Outcome: Insulin Dose Per Body Weight (U/kg) Per Day
Description: Insulin dose in units (U) per body weight in kilograms (kg) per day. Least Squares (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1c, country, sulfonylurea use, time of basal insulin injection, and treatment.
Time Frame: Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline Insulin Dose per Body Weight measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units per kilogram per day (U/kg/day)
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 370 | 372
units per kilogram per day (U/kg/day) | 0.500 (0.03) | 0.479 (0.03)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.393, ANCOVA

10. Secondary Outcome: Insulin Dose (Units)
Description: Units of insulin taken daily. Least Square (LS) means are determined by analysis of covariance (ANCOVA) and adjusted for Baseline HbA1C, country, sulfonylurea use, time of basal insulin injection and treatment.
Time Frame: Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline insulin dose measure; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units per day (U/day)
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 374 | 379
units per day (U/day) | 44.465 (2.62) | 41.015 (2.61)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.185, ANOVA — P-value is for Insulin Dose at Endpoint, up to 24 weeks

11. Secondary Outcome: Percentage of Participants With HbA1c <7 % and HbA1c ≤6.5%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline and 4 weeks and 8 weeks and 12 weeks and 16 weeks and 20 weeks and 24 weeks and Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline HbA1c measure; last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 369 | 375
percentage of participants
  HbA1c- at Baseline < 7.0 % (n=369, 375) | 6.2 | 7.2
  HbA1c- at Baseline ≤ 6.5% (n=369, 375) | 3.5 | 2.4
  HbA1c- at 4 weeks < 7% (n=368, 371) | 16.6 | 15.4
  HbA1c- at 4 week ≤ 6.5%(n=368, 371) | 5.7 | 5.9
  HbA1c- at 8 weeks < 7% (n=359, 358) | 27.0 | 29.9
  HbA1c- at 8 weeks ≤ 6.5% (n=359, 358) | 10.3 | 14.5
  HbA1c- at 12 weeks <7% (n=349, 351) | 39.3 | 43.0
  HbA1c- at 12 weeks ≤ 6.5% (n=349, 351) | 20.3 | 22.8
  HbA1c- at 16 weeks <7% (n=345, 345) | 46.7 | 52.8
  HbA1c- at 16 weeks ≤ 6.5% (n=345, 345) | 24.3 | 28.4
  HbA1c- at 20 weeks < 7% (n=338, 334) | 49.4 | 54.2
  HbA1c- at 20 weeks ≤ 6.5% (n=338, 334) | 26.6 | 32.6
  HbA1c- at 24 weeks < 7% (n=331, 329) | 50.8 | 55.9
  HbA1c- at 24 weeks ≤ 6.5% (n=331, 329) | 27.5 | 32.5
  HbA1c- Endpoint, up to 24 weeks <7% (n=369, 375) | 48.8 | 52.5
  HbA1c- Endpoint, up to 24 weeks ≤ 6.5% (n=369,375) | 26.8 | 30.4
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.661, Chi-squared — P-value is for HbA1c <7% at Baseline
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.394, Chi-squared — P-value is for HbA1c ≤ 6.5% at Baseline
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.688, Chi-squared — P-value is for HbA1c <7% at 4 weeks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p > 0.999, Chi-squared — P-value is for HbA1c ≤ 6.5% at 4 weeks
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.409, Chi-squared — P-value is for HbA1c <7% at 8 weeks
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.090, Chi-squared — P-value is for HbA1c ≤ 6.5% at 8 weeks
Statistical Analysis 7: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.319, Chi-squared — P-value is for HbA1c <7% at 12 weeks
Statistical Analysis 8: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.463, Chi-squared — P-value is for HbA1c ≤6.5% at 12 weeks
Statistical Analysis 9: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.128, Chi-squared — P-value is for HbA1c <7% at 16 weeks
Statistical Analysis 10: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.261, Chi-squared — P-value is for HbA1c ≤6.5% at 16 weeks
Statistical Analysis 11: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.218, Chi-squared — P-value is for HbA1c <7% at 20 weeks
Statistical Analysis 12: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.092, Chi-squared — P-value is for HbA1c ≤6.5% at 20 weeks
Statistical Analysis 13: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.186, Chi-squared — P-value is for HbA1c <7%% at 24 weeks
Statistical Analysis 14: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.174, Chi-squared — P-value is for HbA1c ≤6.5% at 24 weeks
Statistical Analysis 15: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.340, Chi-squared — P-value is for HbA1c <7% at Endpoint, up to 24 weeks
Statistical Analysis 16: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.293, Chi-squared — P-value is for HbA1c ≤6.5% at Endpoint, up to 24 weeks

12. Secondary Outcome: Incidence of Hypoglycemic Events
Description: A hypoglycemic event is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has blood glucose (BG) concentration of ≤70 milligrams/deciliter (mg/dL) even if it was not associated with signs, symptoms, or treatment consistent with current American Diabetes Association (ADA: 2005) guidelines. Severe hypoglycemia is defined as a hypoglycemic event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions (these episodes may be associated with sufficient neuroglycopenia to induce seizure or coma; also, BG measurements may not be available during such an event). Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking.
Time Frame: Baseline and Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline hypoglycemic event measure.
Measure: Number; unit: hypoglycemic events in 24 weeks
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 373 | 376
hypoglycemic events in 24 weeks
  Total Events with BG ≤70 mg/dL | 3564 | 3845
  Severe Events | 7 | 2
  Nocturnal Events with BG ≤70 mg/dL | 1248 | 1386
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.594, Chi-squared — P-value is for Total Hypoglycemic with BG ≤70 mg/dL events
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.462, Chi-squared — P-value is for Nocturnal Hypoglycemic with BG ≤70 mg/dL events

13. Secondary Outcome: Rate Per 30 Days of Hypoglycemic Events
Description: The rate of hypoglycemic events per 30 days between two visits is defined as the total number of events between the visits divided by the actual number of days between the visits, and then multiplied by 30 days. A hypoglycemic event is defined as any time a participant has a blood glucose (BG) level of ≤70 milligrams per deciliter (mg/dL) even if the event was not associated with signs, symptoms, or treatment consistent with current guidelines (American Diabetes Association 2005). Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking. Severe hypoglycemia is defined as a hypoglycemic event requiring assistance of another person to actively administer carbohydrates, glucagons, or other resuscitative actions. Severe Hypoglycemic events may or may not have a reported BG ≤70 mg/dL. These events may be associated with sufficient neuroglycopenia to induce seizure or coma.
Time Frame: Baseline, Endpoint (up to 24 weeks)
Population: All randomized participants who received at 1 dose of study drug with Baseline at least 1 post-Baseline hypoglycemic event.
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 30 days
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 373 | 376
hypoglycemic events per 30 days
  Total Hypoglycemia with BG ≤70 mg/dL | 1.75 (2.00) | 1.83 (2.32)
  Severe Hypoglycemia | 0.00 (0.05) | 0.00 (0.01)
  Nocturnal Hypoglycemia with BG ≤70 mg/dL | 0.61 (0.96) | 0.66 (1.20)
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.995, Wilcoxon (Mann-Whitney) — P-value is for Total Hypoglycemia with BG ≤70 mg/dL events
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.686, Wilcoxon (Mann-Whitney) — P-value is for Nocturnal Hypoglycemia with BG ≤70 mg/dL events

14. Other Pre Specified Outcome: Percentage of Participants With Detectable Insulin Antibody Levels
Time Frame: Baseline and 4 weeks and 12 weeks and 24 weeks and Endpoint (up to 24 weeks) and Baseline to 24 weeks (Overall)
Population: All randomized participants who received at least 1 dose of study drug with Baseline and at least 1 post-Baseline analysis to detect insulin antibodies; last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 365 | 365
percentage of participants
  Baseline (n=365, 365) | 5.5 | 3.6
  4 weeks (n=362, 359) | 7.2 | 3.6
  12 weeks (n= 351, 344) | 7.1 | 6.7
  24 weeks (n=337, 328) | 8.6 | 5.8
  Endpoint, up to 24 weeks (n= 365, 365) | 8.2 | 6.0
  Baseline to 24 weeks (Overall) (n= 365, 365) | 15.3 | 11.0
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.285, Chi-squared — P-value is for Baseline
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.047, Chi-squared — P-value is for 4 weeks
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.882, Chi-squared — P-value is for 12 weeks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.179, Chi-squared — P-value is for 24 weeks
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.314, Chi-squared — P-value is for Endpoint, up to 24 weeks
Statistical Analysis 6: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.100, Chi-squared — P-value is for Baseline to 24 weeks (Overall)

15. Other Pre Specified Outcome: Percentage of Participants With Treatment Emergent Antibody Response (TEAR)
Description: TEAR is defined as an absolute increase of at least 1% in insulin antibody levels (measured in % binding) and at least 30% relative increase from Baseline for participants who are insulin antibody-positive at Baseline, or turning from insulin antibody-negative status at Baseline to antibody-positive during the course of the study following treatment with study drug.
Time Frame: 4 weeks and 12 weeks and 24 weeks and Endpoint (up to 24 weeks) and Baseline to 24 weeks (Overall)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Number analyzed (Participants) | 376 | 380
percentage of participants
  4 weeks (n= 362, 359) | 5.0 | 2.8
  12 weeks (n= 351, 344) | 5.1 | 5.2
  24 weeks (n=337, 328) | 6.2 | 5.2
  Endpoint, up to 24 weeks (n= 365, 365) | 6.0 | 5.5
  Overall (n= 365, 365) | 12.3 | 9.3
Statistical Analysis 1: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.176, Chi-squared — P-value is for 4 weeks
Statistical Analysis 2: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.999, Chi-squared — P-value is for 12 weeks
Statistical Analysis 3: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.618, Chi-squared — P-value is for 24 weeks
Statistical Analysis 4: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p = 0.874, Chi-squared — P-value is for Endpoint (LOCF)
Statistical Analysis 5: Comparison: LY2963016 + OAMs vs Lantus + OAMs; Test type: Superiority or Other; p > 0.233, Chi-squared — P-value is for Overall (Baseline to 24 weeks)

ADVERSE EVENTS:
Arm/Group | LY2963016 + OAMs | Lantus + OAMs
Serious Adverse Events (participants affected / at risk) | 15/376 | 18/380
Other Adverse Events (participants affected / at risk) | 188/376 | 175/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2963016 + OAMs (N=376) | Lantus + OAMs (N=380)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Event resulted in death
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (7) | 3 (3)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Event resulted in death
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/197 (0) | 1/181 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 + OAMs (N=376) | Lantus + OAMs (N=380)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 14 (15)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 8 (10) | 8 (9)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (6)
Oedema peripheral (General disorders) | 5 (5) | 6 (6)
Bronchitis (Infections and infestations) | 5 (5) | 6 (6)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 6 (6)
Influenza (Infections and infestations) | 7 (7) | 11 (12)
Nasopharyngitis (Infections and infestations) | 21 (23) | 22 (27)
Sinusitis (Infections and infestations) | 8 (8) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 19 (21) | 15 (18)
Urinary tract infection (Infections and infestations) | 7 (9) | 7 (7)
Weight increased (Investigations) | 5 (5) | 7 (7)
Abnormal loss of weight (Metabolism and nutrition disorders) | 4 (6) | 3 (4)
Abnormal weight gain (Metabolism and nutrition disorders) | 10 (12) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 10 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6)
Dizziness (Nervous system disorders) | 6 (8) | 5 (7)
Headache (Nervous system disorders) | 8 (8) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (4)
Sinus headache (Nervous system disorders) | 5 (6) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (6)
Hypertension (Vascular disorders) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days